CLINICAL TRIAL: NCT05278663
Title: A Randomized, Double-Blind, Placebo-Controlled, Multi-center, Multiple Ascending Dose Study to Assess the Safety, Tolerability, and Pharmacokinetics of E6742 in Systemic Lupus Erythematosus Patients
Brief Title: A Study to Assess the Safety, Tolerability, and Pharmacokinetics of E6742 in Systemic Lupus Erythematosus Participants
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: E6742-J081-101; jRCT2041210137 (Registry Identifier: jRCT)
Record Dates: First submitted 2022-03-04; First posted 2022-03-14 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-04

CONDITIONS: Lupus Erythematosus, Systemic
Keywords: E6742
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort 1: E6742 100 mg or Placebo (Experimental): Participants will receive E6742 100 milligram (mg) tablet or E6742-matched placebo tablet, orally, twice daily for up to 85 days.
  Interventions: Drug: E6742; Other: Placebo
- Cohort 2: E6742 200 mg or Placebo (Experimental): Participants will receive E6742 200 mg tablets (two tablets of each 100 mg) or E6742-matched placebo tablets, orally, twice daily for up to 85 days.
  Interventions: Drug: E6742; Other: Placebo

INTERVENTIONS:
Drug: E6742 — E6742 tablet.
Other: Placebo — E6742-matching placebo tablet.

SUMMARY:
The primary purpose of the study is to evaluate the safety and tolerability of multiple oral doses of E6742 in participants with systemic lupus erythematosus (SLE).

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female, age greater than or equal to (>=) 18 years and less than or equal to (<=) 75 years at the time of written informed consent
2. Body mass index (BMI) >=15 kilogram per square meter (kg/m^2) and less than (<) 30 kg/m^2 at screening
3. Diagnosed with SLE according to 2019 The European Alliance of Associations for Rheumatology (EULAR)/American College of Rheumatology (ACR) classification criteria, Systemic Lupus International Collaborating Clinics Disease Index (SLICC) classification criteria (2012 version), or 1997 revised ACR classification criteria at least 6 months before the informed consent
4. Meets at least one of the following criteria at screening:

   * Antinuclear antibody positive (>=1:80)
   * Anti-double stranded deoxyribonucleic acid (DNA) antibody positive
   * Anti-smith antibody positive

Exclusion Criteria:

1. Females who are breastfeeding or pregnant at screening or baseline (as documented by a positive beta-human chorionic gonadotropin [ß-hCG] or human chorionic gonadotropin [hCG] test). A separate baseline assessment is required if a negative screening pregnancy test was obtained more than 72 hours before the first dose of study drug
2. Females of childbearing potential who:

   • Within 28 days before study entry, did not use a highly effective method of contraception, which includes any of the following:
   * total abstinence (if it is their preferred and usual lifestyle)
   * an intrauterine device or intrauterine hormone-releasing system (IUS)
   * a contraceptive implant
   * an oral contraceptive (Participant must have been on a stable dose of the same oral contraceptive product for at least 28 days before dosing and must agree to stay on the same dose of the oral contraceptive throughout the study and for 28 days after study drug discontinuation)
   * have a vasectomized partner with confirmed azoospermia
   * Do not agree to use a highly effective method of contraception (as described above) throughout the entire study period and for 28 days after study drug discontinuation
   * Participants on an oral contraceptive must use an additional barrier method throughout the study and for 28 days after study drug discontinuation NOTE: All females will be considered to be of childbearing potential unless they are postmenopausal (amenorrheic for at least 12 consecutive months, in the appropriate age group, and without other known or suspected cause) or have been sterilized surgically (that is, bilateral tubal ligation, total hysterectomy, or bilateral oophorectomy, all with surgery at least 1 month before dosing). Approved or certificated for drugs or medical devices in Japan
3. Males who have not had a successful vasectomy (confirmed azoospermia) if their female partners meet the exclusion criteria above (that is, the female partners are of childbearing potential and are not willing to use a highly effective contraceptive method throughout the study period and for 5 times the half-life of the study drug plus 90 days after study drug discontinuation). No sperm donation is allowed during the study period and for 5 times the half-life of the study drug plus 90 days after study drug discontinuation
4. Any history of surgery that may affect pharmacokinetic (PK) profiles of E6742 (example, hepatectomy, nephrectomy, digestive organ resection) at screening
5. Scheduled for surgery during the study
6. A prolonged QT interval corrected for heart rate using Fridericia's formula (QTcF) (Fridericia method) interval (QTcF greater than [>] 450 millisecond [ms]) as demonstrated by a repeated ECG at screening or baseline. A history of risk factors for torsade de pointes (example, heart failure, hypokalemia, family history of long QT Syndrome) or the use of concomitant medications that prolonged the QTcF interval except for hydroxychloroquine
7. Psychotic disorders or unstable recurrent affective disorders evident by use of antipsychotics within 2 years before screening
8. History of drug or alcohol dependency or abuse within 2 years before screening
9. History of drug allergy or allergy to any investigational product excipients at screening
10. Known to be human immunodeficiency virus (HIV) positive at screening
11. Positive on test at screening for hepatitis B virus surface antigen (HBs antigen), hepatitis B virus surface antibody (HBs antibody), hepatitis B virus core antibody (HBc antibody), hepatitis B virus DNA (HBV DNA), hepatitis C virus antibody (HCV antibody), human T-lymphotrophic virus Type I antibody (HTLV-1 antibody), or syphilis
12. History of clinically significant infections such as latent infectious viruses
13. History of infections requiring hospitalization or intravenous antibiotics, or administration of antiviral drugs, within 4 weeks before the first dose of study drug
14. History of active tuberculosis
15. Any findings indicating a history of tuberculosis on chest X-ray at screening
16. Currently enrolled in another clinical study or used any investigational drug or device within 16 weeks (or 5 half-lives, whichever is longer) before informed consent
17. Received vaccination within 4 weeks before the study treatment (8 weeks before in case of live vaccine)
18. Any history of or concomitant medical condition that in the opinion of the investigators would compromise the participant's ability to safely complete the study
19. Any clinically significant symptom or organ impairment
20. Drug induced lupus erythematosus
21. Active or unstable neuropsychiatric lupus
22. Renal impairment at Screening
23. Systemic autoimmune diseases other than SLE (example, rheumatoid arthritis, Crohn's disease, scleroderma, multiple sclerosis.) that may affect the assessment of SLE pathology
24. History of or complications from malignancy, lymphoma, leukemia, or lymphoproliferative disease (except for basal cell skin cancer, squamous cell skin cancer, and cervical cancer that have been cured by surgical operation)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2022-04-14 (Actual); Primary Completion 2023-09-04 (Actual); Study Completion 2023-09-04 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) | Screening up to 28 days after the last dose of study drug at Day 85 (up to approximately 1 year 5 months)
  Safety assessments will consist of monitoring and recording all adverse events (AEs) and SAEs; laboratory evaluation for hematology, blood chemistry, and urine values; periodic measurement of vital signs and electrocardiograms (ECGs); the performance of physical examinations and chest X-ray test.

SECONDARY OUTCOMES:
Cmax: Maximum Observed Plasma Concentration for E6742 and its Metabolite (ER-001132963) on Days 1 and 15 | Days 1 and 15: 0-6 hours post-dose
Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for E6742 and its Metabolite (ER-001132963) on Days 1 and 15 | Days 1 and 15: 0-6 hours post-dose
AUC(0-6Hours): Area Under the Plasma Concentration Versus Time Curve from Time 0 to 6 Hours for E6742 and its Metabolite (ER-001132963) on Days 1 and 15 | Days 1 and 15: 0-6 hours post-dose

CONTACTS AND LOCATIONS:
Locations (12):
- Japan (12):
  - Chukyo Hospital, Nagoya, Aichi-ken
  - Daido Clinic, Nagoya, Aichi-ken
  - Matsuyama Red Cross Hospital, Matsuyama, Ehime
  - Hospital of the University of Occupational and Environmental Health, Kitakyushu, Fukuoka
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Tohoku University Hospital, Sendai, Miyagi
  - Osaka University Hospital, Suita, Osaka
  - Juntendo University Hospital, Bunkyo-ku, Tokyo
  - St. Luke's International Hospital, Chuo-ku, Tokyo
  - Tokyo Metropolitan Hospital Organization Tokyo Metropolitan Tama Medical Center, Fuchū, Tokyo
  - Center Hospital of the National Center for Global Health and Medicine, Shinjuku-ku, Tokyo
  - National Hospital Organization Kyushu Medical Center, Fukuoka

IPD SHARING:
Plan to Share IPD: Yes
Eisai's data sharing commitment and further information on how to request data can be found on our website http://eisaiclinicaltrials.com/.

REFERENCES:
- [Derived] Tanaka Y, Kumanogoh A, Atsumi T, Ishii T, Tago F, Aoki M, Yamamuro S, Akira S. Safety, pharmacokinetics, biomarker response and efficacy of E6742: a dual antagonist of Toll-like receptors 7 and 8, in a first in patient, randomised, double-blind, phase I/II study in systemic lupus erythematosus. RMD Open. 2024 Sep 17;10(3):e004701. doi: 10.1136/rmdopen-2024-004701. PMID 39289029